CLINICAL TRIAL: NCT03755024
Title: Implementation of WHO Fetal Growth Charts in Assiut,Egypt
Brief Title: WHO Fetal Growth Charts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mina eshak tawfeek khalil, Principal investigator, Assiut University
Other Study IDs: WHOFC
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Fetal Growth Complications
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal group: fetuses with normal growth
  Interventions: Device: ultrasound
- Growth retardation group: fetuses with retarded growth
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — The compulsory ultrasound measurements to be obtained at all visits include the following biometrical parameters:
  * Biparietal diameter
  * Head circumference
  * Abdominal circumference
  * Femur length
  * Humerus length

SUMMARY:
Perinatal mortality and morbidity continue to be major global health challenges strongly associated with prematurity and reduced fetal growth, an issue of further interest given the mounting evidence that fetal growth in general is linked to degrees of risk of common noncommunicable diseases in adulthood. Ultrasound estimation of fetal weight before birth is today very widely used in clinical practice, and, while essential for the identification and management of high-risk pregnancies,the current reference ranges used worldwide are largely based on single populations from a few high-income countries and are therefore of uncertain general applicability.

DETAILED DESCRIPTION:
Against this background, WHO made it a high priority to provide fetal growth charts for estimated fetal weight and common ultrasound biometric measurements intended for worldwide use. WHO study was conducted in 10 countries including Egypt (Assiut).The study showed that fetal growth differs significantly between countries. Growth was to a small extent influenced by maternal age, height, weight, and parity, and by fetal sex. The study suggested that these WHO charts for growth are more suitable for international use than those commonly applied today. However, the differences between countries, with maternal factors, and with fetal sex mean that these growth charts may need to be adjusted for local clinical use to increase their diagnostic and predictive performance. In our setting, we are using the charts built in the ultrasound machines based on studies done in western countries. So, it is prudent now to implement the WHO fetal growth charts in our setting

ELIGIBILITY:
Inclusion Criteria:

* They have body-mass index between 18-30;
* They have a singleton pregnancy;
* Their gestational age at entry is between 8+0 to 12+6 weeks based on last menstrual period.
* They have no history of health, environmental or economic constraints likely to impede fetal growth; need for long-term medication (including fertility treatment); smoking currently or in the previous 6 months; recurrent miscarriage; and any previous baby delivered pre-term (<37 weeks) or with a birth weight <2,500g b. Exclusion criteria:
* Multiple pregnancy
* Congenital fetal malformation (cardiac, cerebral, renal malformations, etc.)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women attending Antenatal care clinic of Women's Health Hospital, Faculty of Medicine, Assiut university.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of fetuses with abnormal fetal growth diagnosed using WHO fetal charts | 8 months
  correlation of fetal growth pattern with neonatal birth weight and outcome